CLINICAL TRIAL: NCT05728840
Title: Virtual-reality Exercises for Alleviating Attention Deficits in Patients with Acquired Brain Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mindmaze SA (Industry)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MFOCUS-1
Record Dates: First submitted 2023-01-26; First posted 2023-02-15 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Attention Disorder
Keywords: stroke; attention; executive functions; virtual reality; neurorehabilitation
MeSH Terms: conditions — Stroke; Cognition Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Rehabilitation intervention group (Experimental): Each participant of the experimental group will undergo an initial cognitive screening (pre-training) and, in addition to their standard of care, they will have 20 additional sessions with the experimental rehabilitation program. Post-treatment cognitive screening will be completed at the end of the program, then 3-4 and 6-12 months later.
  Interventions: Other: Immersive virtual reality gamified cognitive activities
- Dose-match control group (Active Comparator): Each participant of the experimental group will undergo an initial cognitive screening (pre-training) and, in addition to their standard of care, they will have 20 additional sessions of neuropsychological standard sessions. Post-treatment cognitive screening will be completed at the end of the program, then 3-4 and 6-12 months later.
  Interventions: Other: Double neuropsychological standard activities
- Retrospective standard of care group (No Intervention): Each participant of the retrospective group will be included retrospectively if they were hospitalized in the study's sites between 2012 and 2022, and followed standard neuropsychological rehabilitation of attention.

INTERVENTIONS:
Other: Immersive virtual reality gamified cognitive activities — This intervention will include 20 sessions of training with the experimental rehabilitation program using immersive VR cognitive gamified activities, in addition to the standard of care.
  Arms: Rehabilitation intervention group
Other: Double neuropsychological standard activities — This intervention will include 20 sessions of training using a standard neuropsychological rehabilitation program, in addition to the standard of care.
  Arms: Dose-match control group

SUMMARY:
Stroke is the leading cause of long-term disability with an increasing incidence, especially in young adults. Among the cognitive difficulties following brain damage, deficits in attention are frequent and pervasive, affecting between 46% and 92% of stroke survivors. The current project targets patients with acquired brain injury, including stroke, traumatic brain injury, and brain tumor. The main objective of this study is to evaluate the use and the efficacy of a training program targeting attention and executive function difficulties, using gamified and digitized versions in virtual reality of standard cognitive exercises for patients with brain lesions.

DETAILED DESCRIPTION:
Among the cognitive disorders due to stroke, attention impairments are frequent and pervading deficits with a variable incidence ranging from 46% to 92% for attention deficits. Stroke patients may have difficulties to focus, pay attention or attend to more than one stimulus at a time. These deficits are insufficiently addressed in the current standard of care. The proposed study is a three-arm (N=45 per group), double-blind, randomized, and actively controlled study. This study uses immersive virtual reality (VR) based training protocols to address attention and executive dysfunctions in patients with stroke. For each cognitive domain, the solution proposes specific gamified activities, with different levels of difficulty, titrated to the patient's level of impairment, assessed by embedded short assessments. The investigators hypothesize that a daily training using VR-based gamified neuropsychological activities, in addition to standard of care, will decrease attention and executive deficits as much as time-matched daily extra neuropsychological sessions of standard of care. The investigators hypothesize too that delivering such daily extra session of VR-based gamified neuropsychological activities in addition to the standard of care will decrease more attention deficits than the actual regular standard of care dose. The primary outcome will be the change in attentional abilities, measured by standardized tests of attention, before and after 20 sessions of VR-based training for the experimental group and 20 additional neuropsychological are sessions for the dose-match control group. The secondary outcomes will include changes in spatial cognition, attention in activities of daily life, executive functions, influence of the lesions' etiology, impression of our rehabilitation program as a credible treatment, among others.

ELIGIBILITY:
Inclusion Criteria:

* Time from stroke onset < 1 month
* Objective pathological performance on at least one standardized test or subtest on attention during standard neuropsychological evaluation
* Brain injury documented by routine neuroradiological examination (computed tomography or magnetic resonance imaging scan)
* Able to give informed consent as documented by signature
* Age >= 18 years old

Exclusion Criteria:

* Epilepsy
* Inability or contraindications to undergo the investigated intervention
* Major psychiatric co-morbidity
* Major neurocognitive deficits (e.g. dementia)
* Incapacity to discriminate colors
* General cognitive state preventing to understand and perform the tasks
* Decision to not be informed of incidental findings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Test of Attentional Performance (TAP) | Before the intervention (baseline) and after 20 days of training (end of intervention), within 7 weeks from first day of training
  Main deficit of Attention

SECONDARY OUTCOMES:
Test of Attentional Performance (TAP) | Before the intervention (baseline), after 10 days of training (mid-training), 3-4 and 6-12 months after the end of intervention
  Main deficit of Attention
Test of Attentional Performance (TAP) | Before the intervention (baseline), after 20 days of training (end of intervention), 3-4 and 6-12 months after the end of intervention
  Other deficits of attention
Wechsler Memory Scale (WMS-III) | Before the intervention (baseline), after 20 days of training (end of intervention), 3-4 and 6-12 months after the end of intervention
Brief Visuospatial Memory Test (BVMT) | Before the intervention (baseline), after 20 days of training (end of intervention), 3-4 and 6-12 months after the end of intervention
Stroop test | Before the intervention (baseline), after 20 days of training (end of intervention), 3-4 and 6-12 months after the end of intervention
Rating Scale of Attentional Behaviour (RSAB) | Before the intervention (baseline), after 20 days of training (end of intervention), 3-4 and 6-12 months after the end of intervention
Catherine Bergego Scale (CBS) | Before the intervention (baseline), after 20 days of training (end of intervention), 3-4 and 6-12 months after the end of intervention
Stroke impact Scale (SIS) | Before the intervention (baseline), after 20 days of training (end of intervention), 3-4 and 6-12 months after the end of intervention
Far space attention: Hemineglect far space Immersive VR-based task | Before the intervention (baseline), after 20 days of training (end of intervention), 3-4 and 6-12 months after the end of intervention
Response to saliency: Immersive VR-based free-viewing exploration (FVE-VR) task | Before the intervention (baseline), after 20 days of training (end of intervention), 3-4 and 6-12 months after the end of intervention
Credibility/Expectancy Questionnaire (CEQ) | Before the intervention (baseline), after 20 days of training (end of intervention), 3-4 and 6-12 months after the end of intervention
Fatigue: Penner questionnaire | Before the intervention (baseline), after 20 days of training (end of intervention), 3-4 and 6-12 months after the end of intervention
Immersive VR-based attentional performance task | Before the intervention (baseline), after each cycle of 5 days of training, after 20 days of training (end of intervention), 3-4 and 6-12 months after the end of intervention
Defense Automated Neurobehavioral Assessment (DANA) | Before the intervention (baseline), after each cycle of 5 days of training, after 20 days of training (end of intervention), 3-4 and 6-12 months after the end of intervention
User Engagement Scale (UES) | After 20 days of training (end of intervention)
NASA task load index (NASA-TLX) | After 20 days of training (end of intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Crottaz-Herbette, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- University of Lausanne Hospitals, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No